CLINICAL TRIAL: NCT04182360
Title: Carbetocin at Elective Cesarean Deliveries: A Dose-finding Study in Women With Twin Pregnancy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-07
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Postpartum Hemorrhage; Twin
Keywords: Pregnancy; Twins; Postpartum hemorrhage; carbetocin; uterotonic; cesarean delivery
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin

STUDY DESIGN:
Intervention Model Description: Biased coin up-and-down design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Carbetocin 10mcg (Active Comparator): Patient is given 10mcg of carbetocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Carbetocin 20mcg (Active Comparator): Patient is given 20mcg of carbetocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Carbetocin 40mcg (Active Comparator): Patient is given 40mcg of carbetocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Carbetocin 60mcg (Active Comparator): Patient is given 60mcg of carbetocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Carbetocin 80mcg (Active Comparator): Patient is given 80mcg of carbetocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Carbetocin 100mcg (Active Comparator): Patient is given 100mcg of carbetocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — Carbetocin administered intravenously, over 1 minute following delivery of the fetal head.
  Other Names: Duratocin

SUMMARY:
Poor uterine tone after the birth of a baby can cause excess bleeding (called postpartum hemorrhage or PPH). This is a major cause of maternal death worldwide. Uterotonic drugs are used to improve the muscle tone of the uterus after birth, and these are effective at reducing the incidence of PPH. The Society of Obstetricians and Gynecologists of Canada (SOGC) has recommended a single dose of 100 mcg of carbetocin at elective cesarean delivery to promote uterine contraction. In a study performed at Mount Sinai Hospital, the investigators have shown that smaller doses of carbetocin (14.8 mcg) are effective in achieving adequate uterine tone at elective cesarean section.

In these dose-finding studies, women with multiple pregnancies have been excluded. Because women with multiple pregnancy have a higher risk of severe PPH, uterine atony, hysterectomy, prolonged hospital stay and death, it is plausible that a higher dose of carbetocin is required. This question remains unanswered.

The hypothesis is that the ED90 of carbetocin in women with twin pregnancy undergoing elective cesarean delivery under regional anesthesia is greater than 20 mcg but less than 100 mcg.

DETAILED DESCRIPTION:
There is a lack of consensus as to what the optimal uterotonic regime is globally. Furthermore, variability in the international guidelines regarding the choice of first line uterotonic in prevention of PPH adds to the confusion. With the widespread availability of carbetocin in some developed countries, including Canada, the question of which uterotonic to adopt and at which dose becomes even more difficult to ascertain. Studies that have currently been published suggest the ED90 doses of carbetocin and oxytocin provide adequate uterine contraction with possibly fewer side effects associated with the lower dose regimens. There is evidence to suggest that lower doses of both carbetocin provide equivalent uterine contractions with a better side effect profile in patients with a singleton pregnancy. However, there is no clinical dosing data specifically for patients with twin pregnancy. The results of our study will provide guidance to obstetric and anesthetic providers worldwide when deciding what dose of carbetocin to use in women with twin pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Twin Pregnancy
* Elective cesarean delivery under regional anesthesia
* Gestational age ≥ 36 weeks
* No known additional risk factors for postpartum hemorrhage
* Written informed consent to participate in this study

Exclusion Criteria:

* Refusal to give written informed consent
* Allergy or hypersensitivity to oxytocin
* Conditions that may predispose to uterine atony and postpartum hemorrhage such as placenta previa, severe preeclampsia (as defined by SOGC guidelines (25)), polyhydramnios, uterine fibroids, previous history of uterine atony resulting in PPH, or bleeding diathesis and obesity, defined as pre-pregnancy BMI >40
* Hepatic, renal, and vascular disease
* Use of general anesthesia prior to the administration of the study drug

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Uterine tone 2 minutes: questionnaire | 2 minutes
  Uterine tone, defined as satisfactory or unsatisfactory by the obstetrician at 2 minutes after completion of the carbetocin injection.

SECONDARY OUTCOMES:
Uterine tone 5 minutes: questionnaire | 5 minutes
  Uterine tone, defined as satisfactory or unsatisfactory by the obstetrician at 5 minutes after completion of the carbetocin injection.
Additional uterotonics administered | 1 hour
  The drug, dosage and timing of any additional uterotonic medication given during surgery.
Estimated blood loss | 24 hours
  Blood loss will be calculated through the difference in hematocrit values assessed prior to surgery and 24 hours after the cesarean delivery.
Intravenous fluid administered during surgery | 2 hours
  The total volume (ml) of fluid administered from entering the operating room to skin closure.
Hypotension: systolic blood pressure less than 80% of baseline | 2 hours
  Systolic blood pressure < 80% of baseline, from drug administration until end of surgery
Tachycardia: heart rate greater than 130% of baseline | 2 hours
  Heart rate > 130% of baseline, from drug administration until end of surgery
Bradycardia: heart rate less than 70% of baseline | 2 hours
  Heart rate < 70% of baseline or a heart rate < 50bpm, from drug administration until end of surgery
Presence of ventricular tachycardia: ECG | 2 hours
  Presence of ventricular tachycardia as recorded by ECG, from drug administration until end of surgery
Presence of atrial fibrillation: ECG | 2 hours
  Presence of atrial fibrillation as recorded by ECG, from drug administration until end of surgery
Presence of atrial flutter: ECG | 2 hours
  Presence of atrial flutter as recorded by ECG, from drug administration until end of surgery
Presence of nausea: questionnaire | 2 hours
  The presence of nausea and number of episodes, from drug administration until end of surgery, as reported by the patient
Presence of vomiting: questionnaire | 2 hours
  The presence of vomiting and number of episodes, from drug administration until end of surgery
Presence of chest pain: questionnaire | 2 hours
  Any presence of chest pain, from drug administration until end of surgery, as reported by the patient
Presence of shortness of breath: questionnaire | 2 hours
  Any presence of shortness of breath, from drug administration until end of surgery, as reported by the patient
Presence of headache: questionnaire | 2 hours
  Any presence of headache, from drug administration until end of surgery, as reported by the patient
Presence of flushing: questionnaire | 2 hours
  Any presence of flushing, from drug administration until end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No